CLINICAL TRIAL: NCT05440448
Title: Patch-free Occlusion Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Foundation of the Southwest (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Eileen Birch, Senior Research Scientist, Retina Foundation of the Southwest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFSW113A; R01EY022313 (NIH)
Record Dates: First submitted 2022-06-17; First posted 2022-06-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patch-free occlusion therapy (Experimental)
  Interventions: Device: Patch-free occlusion therapy
- Standard-of-care patching with an adhesive patch (Active Comparator)
  Interventions: Device: Adhesive patch

INTERVENTIONS:
Device: Patch-free occlusion therapy — Use of filters in glasses to provide occlusion therapy
  Arms: Patch-free occlusion therapy
Device: Adhesive patch — Standard-of-care occlusion therapy with an adhesive patch
  Arms: Standard-of-care patching with an adhesive patch

SUMMARY:
The purpose of the study is to determine whether a patch-free occlusion therapy leads to better visual outcomes in young children with amblyopia than standard-of-care occlusion therapy with an adhesive patch and whether this is associated with better adherence to the treatment.

DETAILED DESCRIPTION:
This is a single-site randomized clinical trial to compare patch-free occlusion therapy with standard-of-care occlusion therapy with an adhesive patch in young children with amblyopia. Participants will be referred from local pediatric ophthalmologists. Following informed consent, children will complete baseline testing to confirm eligibility and provide pre-treatment measurements of visual acuity, suppression, stereoacuity, motor skills, self-perception, and quality of life. Eligible children will then be randomly allocated to either patch-free occlusion therapy or standard-of-care occlusion therapy with an adhesive patch.

Children will participate in their assigned occlusion therapy at home for 12 weeks (primary outcome). Adherence will be objectively monitored with a Theramon sensor. Vision will be re-assessed at 6 weeks and all tests will be repeated at 12 weeks. The patch-free occlusion group will have an option to continue the patch-free occlusion for and additional 6 or 12 weeks (24 weeks total). The standard-of-care occlusion group will be offered the opportunity to use the patch-free treatment at the 12 week visit through 24 weeks. Children who choose to remain in the study beyond the 12 week primary outcome visit will have vision reassessed at 18 and 24 weeks.

The primary analysis will be a comparison of improvement in amblyopic eye visual acuity (baseline-12 weeks) between the patch-free occlusion group and the standard-of-care patching group. Secondary analyses will include comparisons adherence to each treatment, comparison of the proportion of children in each group with visual acuity ≤0.1 logMAR (recovered) at 6 and 12 weeks visit and 95% CIs (at 6 and 12 weeks), comparisons of changes in extent of suppression, depth of suppression, stereoacuity, motor skills standard scores, self-perception scores, and PedEyeQ domain scores. Associations among hours of treatment, changes in visual acuity, suppression, and stereoacuity, will be explored and modeled for dose-response relationships. In exploratory analyses, we will examine whether there are additional improvements in visual acuity, suppression, or stereoacuity between 12 and 24 weeks for the patch-free group (12, 18, and 24 weeks means and 95% CIs).

ELIGIBILITY:
Inclusion Criteria:

* 3-12 years
* male and female
* strabismic, anisometropic, or combined mechanism amblyopia (visual acuity: 0.3-0.8 logMAR)
* interocular visual acuity difference ≥0.3 logMAR
* wearing glasses (if needed) for a minimum of 8 weeks with no change in visual acuity at 2 visits ≥4 weeks apart
* child's ophthalmologist and family willing to forgo standard patching treatment during the study

Exclusion Criteria:

* Prematurity ≥8 wk
* coexisting ocular or systemic disease
* developmental delay
* myopia > -3.00D

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in amblyopic eye visual acuity measured with a logMAR visual acuity chart | 12 weeks
  change in logMAR relative to baseline

SECONDARY OUTCOMES:
Change in amblyopic eye visual acuity measured with a logMAR visual acuity chart | 6,18, and 24 weeks
  change in logMAR relative to baseline
Adherence to patching or viewing videos with glasses measured with a sensor | 6 and 12 weeks
  cumulative hours of treatment with the patch or glasses used to watch videos objectively monitored with the skin temperature sensitive Theramon sensor
Proportion of children who have recovered | 6 and 12 weeks
  Proportion of children who attain amblyopic eye visual acuity of 0.1 logMAR or better
Change in extent of suppression assessed with W4 test | 6 and 12 weeks
  changes in log deg measure with W4 test
change in stereoacuity assessed with the Randot Preschool Stereoacuity Test | 6 and 12 weeks
  change in log arcsec
Change in motor skills assessed with the Movement Assessment Battery for Children-2 | 12 weeks
  change in Movement Assessment Battery for Children-2 (MABC-2) standard scores relative to baseline (normed and scaled 0-19 for worst to best, with 10=average, 5-6 = "at risk", and <5 = "significant impairment")
Change in self-perception assessed with the Pictorial Scale of Perceived Competence and Social Acceptance for Young Children | 12 weeks
  change in domain scores of the Pictorial Scale of Perceived Competence and Social Acceptance for Young Children (standard scores scaled to range from 0 to 100 for worst to best)
Improvement in quality of life assesses with the Pediatric Eye Questionnaire | 12 weeks
  change in domain scores of the Pediatric Eye Questionnaire (PedEyeQ; Rasch-calibrated and scaled to score from 0 to 100 for worst to best)
Change in depth of suppression assessed with the contrast balance index | 6 and 12 weeks
  change in contrast balance index (ratio of amblyopic eye to fellow eye contrast needed to overcome suppression

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Foundation, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No